CLINICAL TRIAL: NCT07175584
Title: Anal Canal-Sparing Technique During Postoperative Pelvic Radiation Therapy for Cervical Cancer Patients to Reduce Hemorrhoids-related Symptoms: A Multicenter Randomized Clinical Trial
Brief Title: A Clinical Study on Alleviating Hemorrhoids-related Symptoms of Pelvic Radiation Therapy
Acronym: ACS-RT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: RenJi Hospital (Other); Suzhou Municipal Hospital (Other); Changzhou Cancer Hospital of Soochow University (Other); The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, Yong Liu, Professor, M.D., Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHGH_IIT2025-070
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hemorrhoidal Disease; Cervical Cancer Radiation Complications
Keywords: cervical cancer; hemorrhoidal disease; pelvic radiation therapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anal Canal-Sparing Arm (Experimental): Participants will receive pelvic radiation therapy using anal canal-sparing techniques. There will be 150 participants enrolled.
  Interventions: Radiation: anal canal-sparing techniques
- Conventional Radiation therapy Arm (No Intervention): Participants will receive pelvic radiation therapy using standard techniques. There will be 150 participants enrolled.

INTERVENTIONS:
Radiation: anal canal-sparing techniques — To contour anal canal and rectum separately and deliver different doses as two single OARs in pelvic radiation therapy planning.
  Arms: Anal Canal-Sparing Arm

SUMMARY:
The goal of this clinical trial is to reduce the acute hemorrhoids-related symptoms for cervical cancer patients with hemorrhoids who need postoperative pelvic radiation therapy, including prolapse, local burning, bleeding, perianal pain, and other perianal discomforts.

The main questions it aims to answer are:

Will anal canal-sparing technique improve the quality of life for cervical cancer patients with hemorrhoids during pelvic radiation therapy? Will the radiation dose exposure to anal canal be reduced through anal canal-sparing technique?

Researchers will compare the aggravation of radiation-induced hemorrhoids-related symptoms occurring from the initiation of pelvic radiation therapy until 4 weeks after its completion. Conventional postoperative treatment regimens will not be changed and researchers will only reduce the irradiated dose to anal canal which should be protected during pelvic radiation therapy.

Participants will be randomly assigned with equal probability (1:1 ratio) to either: control group (conventional postoperative pelvic radiation therapy) and intervention group (anal canal-sparing pelvic radiation therapy), in either combined with brachytherapy or not. Following randomization, participants will not be informed of their group assignment until completion of the follow-up period.

Notice: The treatment efficacy will not be compromised by group assignment. No additional treatment-related adverse effects will occur due to study participation. The intervention group may potentially mitigate radiotherapy-induced adverse effects.

DETAILED DESCRIPTION:
Radiation therapy (RT) is a main treatment method to improves local control and overall survival for cervical cancer patients with high-risk factors. External beam radiation therapy (EBRT) is particularly important, which plays a crucial role for patients either after surgery or for those ineligible for surgery. In intensity-modulated radiation therapy (IMRT) era, 90-95% of patients with pelvic malignancies, including gynecological tumors, still develop varying degrees of radiation-induced intestinal injury. Radiation-induced rectal injury (RRI) is still one of the most common complications of radiation to the pelvis, but which is also the most difficult to treat.

However, whether from the symptoms or the pelvic radiation therapy plans, current studies on RRI generally combine the rectum and anal canal. Therefore, the so-called "Radiation-induced rectal injury" is not purely "rectal injury," but includes "radiation-induced rectal and anal canal injury." In addition, the radiation of perianal muscles can also lead to symptoms related to the rectum during pelvic radiation therapy. According to current contouring guidelines, whether for gynecologic tumors or other pelvic malignancies, the anal canal is regarded together with the rectum as the same organ at risk (OAR) when formulating pelvic EBRT plans, and a unified dose constraint standard is applied. The anal canal and its surrounding muscles are not assessed separately.

The tolerance dose of the rectum is generally considered to be around 50 Gy, however, anal canal-related symptoms may occur at lower doses, particularly in patients with a history of hemorrhoids. During the early phase of radiotherapy, hemorrhoids-associated symptoms such as perianal pain, hemorrhoidal prolapse, rectal bleeding, and perianal skin breakdown may occur. These symptoms are more likely attributable to the aggravation of pre-existing hemorrhoids rather than radiation-induced rectal injury. Hemorrhoidal disease (HD) is one of the most common gastrointestinal disorder managed in outpatient clinics. Although it is not a life-threatening condition, it can persistently and severely impact quality of life and increase the healthcare burden on society.

Anal canal toxicity should not be a neglected side-effect of pelvic radiation therapy, and greater attention need to be paid to the occurrence of acute hemorrhoid-related symptoms, particularly for cervical cancer patients with hemorrhoids. The investigators tried to develop anal canal-sparing technique to reduce the irradiated dose to anal canal for cervical cancer patients with hemorrhoids who needed postoperative pelvic radiation therapy.

Minimizing acute toxic effects is of considerable importance to improve quality of life because it has been correlated with late toxic effects in patients with pelvic radiation therapy. Herein, the investigators design a multicenter, double-blind randomized controlled trial in which cervical cancer patients with hemorrhoids were randomly assigned to receive anal canal-sparing or standard postoperative pelvic radiation therapy, in either combined with brachytherapy or not.

The primary objectives are to compare the incidence of hemorrhoidal symptom and differences in quality of life (QoL) scores during radiotherapy between the two arms. Concurrently, the study will explore the practical implementation methodology of the anal canal-sparing technique.

ELIGIBILITY:
Inclusion Criteria:

* Treated with hysterectomy (including total abdominal hysterectomy, vaginal hysterectomy, radical hysterectomy, or laparoscopically assisted vaginal hysterectomy) within 6 weeks prior to study initiation.
* Histologically proven diagnosis of cervical carcinoma, including squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma.
* Requirement for postoperative adjuvant concurrent chemoradiotherapy (CCRT).
* Age > 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* History of hemorrhoids prior to radiotherapy, with no hemorrhoid-related symptoms for at least 4 weeks before radiation therapy initiation.
* Abdominal/pelvic MRI, chest CT, or PET-CT performed before surgery or study enrollment to confirm staging and exclude patients with distant metastasis.
* Adequate bone marrow, renal, and hepatic function.
* Agreement to undergo anal canal MRI before radiation therapy initiation.
* Patient must provide study-specific informed consent form (ICF) prior to study entry.

Exclusion Criteria:

* Cervical cancer patients who do not meet the criteria for adjuvant radiation therapy.
* Without a confirmed history of hemorrhoids.
* Patients contraindicated for MRI (e.g., due to incompatible metallic implants, claustrophobic syndrome, or other contraindications).
* Patients who refuse to undergo anal canal MRI.
* Patients with radiographically visible residual disease post-surgery requiring boost during the pelvic EBRT.
* History of other malignancies.
* Prior pelvic radiotherapy resulting in overlapping radiation fields.
* History of allergic reaction to platinum-based chemotherapy agents.
* Severe and/or active comorbidities precluding tolerance of concurrent chemoradiotherapy.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2027-09-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of radiation-induced hemorrhoid-related symptoms | From the initiation of pelvic radiation therapy (including BT) until 4 weeks after its completion.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT07175584/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT07175584/ICF_001.pdf